CLINICAL TRIAL: NCT00489918
Title: A Dose Ranging Study of the Effects of Macroflux® PTH Compared With Macroflux® Placebo and FORTEO® in Postmenopausal Women With Osteoporosis
Brief Title: Dose Ranging Study - Macroflux Parathyroid Hormone (PTH) in Postmenopausal Women With Osteoporosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zosano Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP-2006-001
Record Dates: First submitted 2007-06-19; First posted 2007-06-21 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Parathyroid Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Macroflux® placebo (Placebo Comparator): Macroflux® placebo patch
  Interventions: Drug: teriparatide
- Macroflux® 20 mcg (Experimental): Macroflux® 20 mcg patch
  Interventions: Drug: teriparatide
- Macroflux® 30 mcg (Experimental): Macroflux® 30 mcg patch
  Interventions: Drug: teriparatide
- Macroflux® 40 mcg (Experimental): Macroflux® 40 mcg patch
  Interventions: Drug: teriparatide
- FORTEO® (Active Comparator): FORTEO® 20 mcg injection
  Interventions: Drug: teriparatide

INTERVENTIONS:
Drug: teriparatide — Macroflux® patch applied to the abdomen for 30 minutes daily
  Other Names: PTH(1-34)
  Arms: Macroflux® 20 mcg; Macroflux® 30 mcg; Macroflux® 40 mcg; Macroflux® placebo
Drug: teriparatide — FORTEO® injection administered subcutaneously (SC) either to the abdomen or thigh
  Other Names: FORTEO®
  Arms: FORTEO®

SUMMARY:
A Multi-center study to determine effects of various doses of Macroflux Parathryroid Hormone (PTH) in women with osteoporosis

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women age 50 years or older
* At least three lumbar vertebrae (L1-L4) must be evaluable by dual energy x-ray absorptiometry (DXA) for bone mineral densitometry that is, without fracture or significant degenerative disease, as determined by the central imaging facility
* Have osteoporosis defined as: Either a T-score of ≤ -2.5 at the lumbar spine, femoral neck, or total hip, AND a T-score of at least < -1.0 at the lumbar spine; or A T-score of ≤ -2.0 at the lumbar spine, femoral neck, or total hip, AND at least one vertebral fracture;

Exclusion Criteria:

* Active hepatitis;
* Active pancreatitis;
* Unstable cardiac disease;
* Unstable pulmonary disease;
* Celiac disease;
* Hyper- or hypo-parathyroidism;
* Hyperthyroidism;
* Cushing's disease;
* Osteomalacia;
* Paget's disease;
* Osteogenesis imperfecta;
* Known blood disorders;
* History of kidney stones;
* Impaired renal function;
* Autoimmune diseases;
* Bone metastases or a history of skeletal malignancies;
* Cancer history that includes any cancer within the previous 5 years, with the exception of squamous or basal cell carcinoma of the skin in which the lesions were fully resected with clear margins described in a written report by a pathologist, and the patient has had no recurrence of lesions for at least 1 year from the time of original resection;
* Any condition or disease that may interfere with the ability to have or the evaluation of a DXA scan, for example, severe osteoarthritis of the spine, spinal fusion, pedicle screws, history of vertebroplasty, or degenerative disease that results in insufficient number of evaluable lumbar vertebrae, or >1 lumbar vertebral fracture in L1-L4;
* More than 4 vertebral fractures in T4-L4;
* Bilateral hip replacements;
* Use of fluoride (e.g. fluoride therapy for osteoporosis) or strontium at any time;
* Have received methotrexate or immunomodulatory agents with antiproliferative activity;
* With known dermatological disorders that would interfere with the study procedures or assessments, or with a history of contact dermatitis;
* With known allergy or sensitivity to tapes, adhesives, PTH, teriparatide or its analogs, or components of the Macroflux® systems;
* Who, in the opinion of the investigator, should not participate in the study, or may not be capable of following the study schedule for any reason; and
* Unwillingness or inability to abide by the requirements of the study.
* Have received any intravenous (IV) administered bisphosphonates in the past 24 months, or >2 doses of IV administered bisphosphonates total;
* Use of oral bisphosphonates before randomization, including investigational bisphosphonates, unless: <6 months of treatment and off for 6 months, or 6-12 months of treatment and off for 2 years, or >12 months of treatment and off for 5 years;

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten von Stein, MD, Ph.D, Study Director — Zosano Pharma Corporation

REFERENCES:
- [Derived] Cosman F, Lane NE, Bolognese MA, Zanchetta JR, Garcia-Hernandez PA, Sees K, Matriano JA, Gaumer K, Daddona PE. Effect of transdermal teriparatide administration on bone mineral density in postmenopausal women. J Clin Endocrinol Metab. 2010 Jan;95(1):151-8. doi: 10.1210/jc.2009-0358. Epub 2009 Oct 26. PMID 19858319

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO®
Started | 33 | 34 | 32 | 33 | 33
Completed | 31 | 32 | 28 | 32 | 32
Not Completed | 2 | 2 | 4 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Postmenopausal women with osteoporosis
Groups:
- Total: Total of all reporting groups
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO® | Total
Number analyzed (Participants) | 33 | 34 | 32 | 33 | 33 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (7.1) | 64.1 (7.5) | 63.6 (5.8) | 64.6 (7.3) | 63.2 (6.8) | 64.06 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 32 | 33 | 33 | 165
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 4 | 9 | 10 | 14 | 8 | 45
  Hispanic | 29 | 25 | 22 | 19 | 24 | 119
  Asian | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Lumbar Spine Bone Mineral Density (BMD): Baseline to Week 24
Description: Percent Change in Lumbar Spine Bone Mineral Density (BMD) from Baseline to Week 24
Time Frame: 24 weeks
Population: Intent to treat (ITT)/Safety Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO®
Number analyzed (Participants) | 33 | 34 | 32 | 33 | 33
percent change | -0.33 (3.467) | 2.96 (3.524) | 3.47 (3.575) | 4.97 (4.114) | 3.55 (3.730)

2. Secondary Outcome: Percent Change in Lumbar Spine Bone Mineral Density: Baseline to Week 12
Description: Percent Change in Lumbar Spine Bone Mineral Density from Baseline to Week 12
Time Frame: 12 weeks
Population: ITT/Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO®
Number analyzed (Participants) | 33 | 34 | 32 | 33 | 33
Percent change | 0.97 (3.312) | 1.55 (2.606) | 2.04 (3.277) | 2.5 (2.86) | 2.81 (2.771)

3. Secondary Outcome: Absolute Change in Lumbar Spine BMD: Baseline to Week 12
Description: Absolute Change in Lumbar Spine BMD from Baseline to Week 12
Time Frame: 12 weeks
Population: ITT/Safety Population
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO®
Number analyzed (Participants) | 33 | 34 | 32 | 33 | 33
g/cm^2 | 0.007 (0.0234) | 0.011 (0.0191) | 0.014 (0.0238) | 0.017 (0.0285) | 0.021 (0.0201)

4. Secondary Outcome: Percent Change in Total Hip Bone Mineral Density: Baseline to Week 24
Description: Percent Change in Total Hip Bone Mineral Density from Baseline to Week 24
Time Frame: 24 Weeks
Population: ITT/Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO®
Number analyzed (Participants) | 33 | 34 | 32 | 33 | 33
Percent change | -0.634 (1.9719) | 0.138 (2.0386) | 0.553 (2.3694) | 1.331 (2.1111) | 0.094 (2.6194)

5. Secondary Outcome: Percent Change in Femoral Neck BMD: Baseline to Week 24
Description: Percent Change in Femoral Neck BMD from Baseline to Week 24
Time Frame: 24 Weeks
Population: ITT/Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO®
Number analyzed (Participants) | 33 | 34 | 32 | 33 | 33
Percent change | 0.172 (3.3432) | 0.949 (3.2975) | 0.599 (2.6127) | 0.750 (2.6132) | -0.012 (3.6600)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Macroflux® Placebo | Macroflux® 20 mcg | Macroflux® 30 mcg | Macroflux® 40 mcg | FORTEO®
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/34 | 0/32 | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 29/33 | 32/34 | 31/32 | 30/33 | 23/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macroflux® Placebo (N=33) | Macroflux® 20 mcg (N=34) | Macroflux® 30 mcg (N=32) | Macroflux® 40 mcg (N=33) | FORTEO® (N=33)
Subdural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Dehydration due to gastroenterocolitis
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Macroflux® Placebo (N=33) | Macroflux® 20 mcg (N=34) | Macroflux® 30 mcg (N=32) | Macroflux® 40 mcg (N=33) | FORTEO® (N=33)
Application site erythema (Skin and subcutaneous tissue disorders) | 13 | 13 | 15 | 13 | 1
Application site discolorations (Skin and subcutaneous tissue disorders) | 3 | 11 | 11 | 7 | 0
Application site bruising (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 2 | 0
Application site bleeding (Skin and subcutaneous tissue disorders) | 0 | 8 | 14 | 1 | 0
Application site edema (Skin and subcutaneous tissue disorders) | 1 | 2 | 3 | 1 | 0
Edema peripheral (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 1 | 4 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 2 | 1
Influenza (Infections and infestations) | 2 | 2 | 2 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 2
Bronchitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 4 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 4 | 0 | 4 | 6
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 3 | 2 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 5 | 4 | 3 | 4
Dizziness (Nervous system disorders) | 0 | 3 | 1 | 1 | 0
Hypertension (Vascular disorders) | 2 | 1 | 0 | 2 | 0
Hypercalciuria (Renal and urinary disorders) | 2 | 4 | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No